CLINICAL TRIAL: NCT06703190
Title: Estimated Vaccine Effectiveness (VE) and Durability of Pfizer/BioNTech 2024-2025 COVID-19 (Coronavirus Disease 2019) Vaccine
Brief Title: Estimated Vaccine Effectiveness and Durability of Pfizer/BioNTech 2024-2025 COVID-19 Vaccine
Acronym: C4591068
Status: Terminated | Type: Observational
Why Stopped: This secondary data analysis of symptomatic CVS MinuteClinics patients testing for SARS-CoV-2 was terminated due to incomplete data on KP.2 vaccination status (exposure). Termination was not based on any safety concerns or regulatory requirements.
Sponsor: Pfizer (Industry)
Collaborators: CVS Caremark (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591068; NCT06703190 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-11-22; First posted 2024-11-25 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19; Omicron; KP.2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants testing positive for COVID-19 (i.e., cases): Participants testing positive for SARS-CoV-2 infection by RAT at a CVS MinuteClinic and reporting at least one COVID-19 symptom
  Interventions: Biological: Pfizer-BioNTech BNT162b2 COVID-19 Vaccinated; Biological: Not vaccinated with 2024-2025 formulated COVID-19 vaccine
- Participants testing negative for COVID-19 (i.e. negative controls): Participants testing negative for SARS-CoV-2 by RAT at a CVS MinuteClinic and reporting at least one COVID-19 symptom
  Interventions: Biological: Pfizer-BioNTech BNT162b2 COVID-19 Vaccinated; Biological: Not vaccinated with 2024-2025 formulated COVID-19 vaccine

INTERVENTIONS:
Biological: Pfizer-BioNTech BNT162b2 COVID-19 Vaccinated — Non-interventional observed exposure of the receipt of the Pfizer-BioNTech BNT162b2 COVID-19 vaccine (2024-2025 formulation) ≥14 days before testing for SARS-CoV-2
  Other Names: Exposed
Biological: Not vaccinated with 2024-2025 formulated COVID-19 vaccine — The reference group will be no receipt of the Pfizer-BioNTech BNT162b2 COVID-19 vaccine (2024-2025 formulation), or any other 2024-2025 formulated COVID-19 vaccine, ≥14 days before testing for SARS-CoV-2.
  Other Names: Unexposed

SUMMARY:
This study is a retrospective case control analysis on the real-world effectiveness of the Pfizer-BioNTech BNT162b2 vaccine (2024-2025 formulation) against symptomatic SARS-CoV-2 infection among CVS MinuteClinic patients testing for SARS-CoV-2, across different age groups, during periods of various variant circulation, and by months since receipt of vaccine dose.

DETAILED DESCRIPTION:
Background:

Omicron and its sublineages have comprised of the majority of SARS-CoV-2 genomes sequenced by the Centers for Disease Control and Prevention (CDC) since December 2021. KP.2 was first identified as a circulating variant under monitoring (VUM) by the World Health Organization in March 2024. FLiRT-mutated subvariants (including KP.2 and recent FluQE-mutated subvariants) have been the predominant variants sequenced in the US throughout 2024. FLiRT-mutated sub-lineages are antigenically distant from prior circulating SARS-CoV-2 lineages, including Omicron XBB, Omicron BA.4/BA.5 and the original SARS-CoV-2 wild-type strain. While Omicron XBB-adapted vaccines provide some protection against a range of outcomes from FLiRT-mutated-related COVID-19, evidence suggests that vaccines better matched to currently circulating sub-lineages can help further improve protection against symptomatic disease and severe COVID-19. Following guidance from regulatory authorities on the requirements for strain changes, Pfizer/BioNTech filed data showing that the FLiRT-mutated-adapted (KP.2) monovalent COVID-19 vaccine generates improved responses against circulating sublineages, compared to the 2023-2024 Omicron XBB-adapted COVID-19 vaccine. On June 27, 2024, the Advisory Committee on Immunization Practices recommended an updated 2024-2025 COVID-19 vaccine for all persons aged ≥6 months, regardless of prior vaccination history. On August 22nd 2024, FDA approved the KP.2 strain COVID-19 vaccine (2024-2025 Formula) for those aged >12 years ages and authorized its use in those 6 months through 11 years of age.

Research Question:

What is the real-world effectiveness of the Pfizer/BioNTech 2024-2025 formulation of the COVID-19 vaccine against symptomatic COVID-19, across different age groups, during periods when different subvariants are circulating, and by months since receipt of the 2024-2025 formulated COVID-19 vaccine dose?

Research Methods:

Population: In collaboration with CVS, Pfizer will conduct a retrospective study to analyze patients tested for SARS-CoV-2 on or after September 5th, 2024, which corresponds with 14 days following FDA approval of the 2024-2025 updated COVID-19 vaccine. CVS will leverage CVS MinuteClinic data on patients ≥5 years of age who are testing for SARS-CoV-2 to evaluate the effectiveness of the 2024-2025 Pfizer/BioNTech COVID-19 vaccine formulation against symptomatic SARS-CoV-2 infection.

Exposure: The exposure of interest will be receipt of the Pfizer-BioNTech BNT162b2 COVID-19 vaccine (2024-2025 formulation) ≥14 days before testing for SARS-CoV-2. The reference group for the overall VE will be no receipt of the Pfizer-BioNTech BNT162b2 COVID-19 vaccine (2024-2025 formulation) or any other 2024-2025 formulated COVID-19 vaccine regardless of prior vaccination history.

Outcome: Cases will be defined as patients testing positive for SARS-CoV-2 infection by RAT at a CVS MinuteClinic and reporting at least one COVID-19 symptom. Controls will be defined as participants testing negative for SARS-CoV-2 by RAT at a CVS MinuteClinic and reporting at least one COVID-19 symptom during the same period.

Calculation: Estimated vaccine effectiveness will be calculated as 1 minus the odds ratio from logistic regression models multiplied by 100.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. MinuteClinic Patients (at least 5 years of age) testing for SARS-CoV-2 on or after September 5th 2024 (at least 14 days after FDA approval of the updated 2024-2025 COVID-19 vaccine formulation); AND
2. At least one symptom reported on the ICATT questionnaire; AND
3. No evidence of a positive SARS-CoV-2 test or COVID-19 diagnosis (or COVID-19 antiviral medications picked up at CVS) within the prior 90 days; AND
4. Vaccine status reported on the ICATT questionnaire and/or ability to confirm receipt of the 2024-2025 formulated COVID-19 vaccine via CVS or Aetna records; AND

   1. Received Pfizer-BioNTech BNT162b2 COVID-19 vaccine (2024-2025 formulation); OR
   2. Did not receive any 2024-2025 formulated COVID-19 vaccine (regardless of manufacturer)

Exclusion Criteria:

Patients meeting any of the following criteria will NOT be included in the study:

1. Those testing at drive-thru locations;
2. Those who tested but are without a completed ICATT questionnaire
3. Those with invalid test results
4. Those not reporting any symptoms
5. Those who received a 2024-2025 formulated COVID-19 vaccine other than from Pfizer/BioNTech (confirmed via a combination of patient- or provider-report and validation against CVS or Aetna vaccination data).
6. Those who received a 2024-2025 formulated COVID-19 vaccine <14 days prior to the test date.
7. Those who reported "prefer not to answer" for vaccination history (and no evidence from CVS vaccination or Aetna data that the patient had received the Pfizer/BioNTech COVID-19 vaccine [2024-2025 formulation]).
8. Those who tested multiple times during the study period.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include retrospectively gathered data from those testing for SARS-CoV-2 at a CVS MinuteClinic
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Number of Pfizer/BioNTech 2024-2025 formulation vaccinated patients who test positive for SARS-CoV-2 ≥14 days after receipt of vaccine | September 2024 - April 2025
  Exposed Cases will be defined as patients testing positive for SARS-CoV-2 infection by RAT at a CVS MinuteClinic and reporting at least one COVID-19 symptom and were vaccinated with the 2024-2025 formulation of the Pfizer/BioNTech vaccine ≥14 days prior to testing.
Number of COVID-19 2024-2025 formulation unvaccinated patients who test positive for SARS-CoV-2 | September 2024 - April 2025
  Unexposed Cases will be defined as patients testing positive for SARS-CoV-2 infection by RAT at a CVS MinuteClinic and reporting at least one COVID-19 symptom and were not vaccinated with any 2024-2025 formulation of COVID-19 vaccine ≥14 days prior to testing.
Number of Pfizer/BioNTech 2024-2025 formulation vaccinated patients who test negative for SARS-CoV-2 ≥14 days after receipt of vaccine | September 2024 - April 2025
  Exposed Controls will be defined as patients testing negative for SARS-CoV-2 infection by RAT at a CVS MinuteClinic and reporting at least one COVID-19 symptom and were vaccinated with the 2024-2025 formulation of the Pfizer/BioNTech vaccine ≥14 days prior to testing.
Number of COVID-19 2024-2025 formulation unvaccinated patients who test negative for SARS-CoV-2 | September 2024 - April 2025
  Unexposed Controls will be defined as patients testing negative for SARS-CoV-2 infection by RAT at a CVS MinuteClinic and reporting at least one COVID-19 symptom and were not vaccinated with any 2024-2025 formulation of COVID-19 vaccine ≥14 days prior to testing.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591068